CLINICAL TRIAL: NCT00295880
Title: A Phase I/II Study of Double Unit Umbilical Cord Blood (UCB) Transplantation Utilizing Graft Administration Via Intra-Bone Marrow Injection (Companion Protocol to MT2000-25)
Brief Title: Donor Umbilical Cord Blood Transplant By Injection Into the Bone Marrow in Treating Patients With Hematologic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Time to engraftment would not be improved compared to historical controls.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004LS072; UMN-MT2004-26 (Other: Blood and Bone Marrow Transplant Program); UMN-0412M65789 (Other: IRB at University of Minnesota)
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Results first posted 2009-09-03 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Myeloproliferative Disorders; Leukemia; Lymphoma; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia in remission; adult acute myeloid leukemia; childhood acute myeloid leukemia in remission; secondary acute myeloid leukemia; accelerated phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; refractory anemia with excess blasts; de novo myelodysplastic syndromes; myelodysplastic syndromes; adult diffuse large cell lymphoma; adult diffuse mixed cell lymphoma; adult diffuse small cleaved cell lymphoma; adult lymphoblastic lymphoma; grade 3 follicular lymphoma; mantle cell lymphoma; childhood large cell lymphoma; childhood lymphoblastic lymphoma; adult acute lymphoblastic leukemia; acute lymphoblastic leukemia; refractory anemia; refractory cytopenia; childhood acute myeloid leukemia; adult immunoblastic large cell lymphoma; blastic phase chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic neutrophilic leukemia; childhood small noncleaved cell lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Anemia, Refractory, with Excess of Blasts; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Dendritic Cell Sarcoma, Interdigitating; Anemia, Refractory; Cytopenia; Lymphoma, Large-Cell, Immunoblastic; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Burkitt Lymphoma | interventions — Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplant Patients (Experimental): Patients receiving umbilical cord blood transplantation.
  Interventions: Procedure: umbilical cord blood transplantation

INTERVENTIONS:
Procedure: umbilical cord blood transplantation — The graft will be given by slow injection into each posterior iliac crest.
  Other Names: UCBT

SUMMARY:
Rationale: Giving chemotherapy and total-body irradiation before a donor umbilical cord blood transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from the donor's umbilical cord blood are injected into the patient's bone marrow they may help make stem cells, red blood cells, white blood cells, and platelets.

Purpose: This phase I/II trial is studying the side effects of donor umbilical cord blood transplant when given directly into the bone marrow and to see how well it works in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
Objectives:

Primary

* Determine the safety, in terms of infusional toxicity, of myeloablative unrelated donor double-unit umbilical cord blood (UCB) transplantation via intra-bone marrow injection (IBMI) in patients with advanced or high-risk hematologic malignancy.
* Determine whether treatment with this regimen improves the time to neutrophil engraftment (compared to historical controls) in these patients.

Secondary

* Determine the incidence of sustained donor engraftment in patients treated with this regimen.
* Determine the relative contribution of each UCB unit to initial and sustained donor engraftment in these patients.
* Determine the incidence of grade II-IV and grade III-IV acute graft-vs-host disease (GVHD) and chronic GVHD in patients treated with this regimen.
* Determine the incidence of day 100 and 180 transplant-related mortality in patients treated with this regimen.
* Determine the probability of survival at 100 days and 1 year post-transplantation in these patients.

Outline: This is a nonrandomized study.

Patients receive a myeloablative conditioning regimen. Patients also receive immunosuppression, growth factor, and supportive care as in protocol MT2005-10 (NCT00309842).

Patients receive 2 units of donor umbilical cord blood (UCB) by intra-bone marrow injection (IBMI) over 10 minutes each on day 0. If the IBMI procedure is not possible, then the UCB units are given intravenously (IV.)

After completion of study therapy, patients are followed periodically for 5 years.

Projected Accrual: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia (AML): high risk CR1
* Acute lymphocytic leukemia (ALL): high risk CR1 [t(9;22), t (1:19), t(4;11) or other MLL rearrangements] or > 1 cycle to obtain CR; CR2+. All patients must be in CR as defined by hematological recovery, AND <5% blasts by light microscopy within the bone marrow with a cellularity of ≥15%.
* Chronic myelogenous leukemia (CML) excluding refractory blast crisis. To be eligible in first chronic phase (CP1) patient must have failed or be intolerant to imatinib mesylate.
* Myelodysplasia (MDS) IPSS Int-2 or High risk (i.e. RAEB, RAEBt) or refractory anemia with severe pancytopenia or high risk cytogenetics.
* Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), marginal zone B-cell lymphoma or follicular lymphoma that have progressed after at least two prior therapies. Patients with bulky disease (nodal mass greater than 5 cm).
* Lymphoplasmacytic lymphoma, mantle-cell lymphoma, prolymphocytic leukemia are eligible after initial therapy in CR1+ or PR1+.
* Large cell NHL > CR2/> PR2. Patients in CR2/PR2 with initial short remission (<6 months) are eligible.
* Lymphoblastic lymphoma.
* Multiple myeloma beyond PR2.
* Karnofsky performance status (PS) 90-100% (adults)
* Lansky PS 50-100% (children)
* Acceptable organ function

Exclusion Criteria:

* Active infection at time of transplantation
* History of HIV infection
* Pregnant or breast feeding.
* Chemotherapy refractory large cell and high grade NHL (ie progressive disease after > 2 salvage regimens)
* Extensive prior therapy including > 12 months alkylator therapy or > 6 months alkylator therapy with extensive radiation.
* Diffuse myelofibrosis of BM (bone marrow) (any severity) regardless of primary diagnosis (focal fibrosis acceptable provided it involves < 20% of BM volume).
* History of pelvic irradiation.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2005-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Wagner, MD, Study Chair — Masonic Cancer Center, University of Minnesota

REFERENCES:
- [Result] Brunstein CG, Barker JN, Weisdorf DJ, Defor TE, McKenna D, Chong SY, Miller JS, McGlave PB, Wagner JE. Intra-BM injection to enhance engraftment after myeloablative umbilical cord blood transplantation with two partially HLA-matched units. Bone Marrow Transplant. 2009 Jun;43(12):935-40. doi: 10.1038/bmt.2008.417. Epub 2009 Jan 12. PMID 19139736

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients are recruited from within the Department of Blood and Marrow Transplant Program. (Patients will be co-enrolled on study MT2005-10 (NCT00309842). Eligibility for this study are identical to MT2005-10.)
Groups:
- Umbilical Cord Blood Transplant Patients: Patients with high-risk hematologic malignancy transplanted with umbilical cord blood via direct marrow injection.
Period: Overall Study
Arm/Group | Umbilical Cord Blood Transplant Patients
Started | 12
Completed | 10
Not Completed | 2
Not completed — IBMI unit could not be volume reduced | 1
Not completed — Unit randomization did not occur | 1

BASELINE CHARACTERISTICS:
Arm/Group | Umbilical Cord Blood Transplant Patients
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Median Number of Days to Neutrophil Engraftment
Description: Number of days to neutrophil recovery observed in recipients of two umbilical cord blood units (UCB)administered i.v. Neutrophil recovery is defined as first of 3 consecutive days with ANC (absolute neutrophil count) greater than or equal to 500/ul.
Time Frame: Daily through Day 60 post transplant
Measure: Median (Full Range); unit: Days
Arm/Group | Umbilical Cord Blood Transplant Patients
Number analyzed (Participants) | 10
Days | 21 [17 to 49]

2. Secondary Outcome: Number of Patients Achieving Neutrophil Recovery
Description: Number of patients with sustained neutrophil recovery with chimerism (evidence of engraftment of both cord blood transplants) at 6 months.
Time Frame: 6 months
Population: Patients who completed treatment.
Measure: Number; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant Patients
Number analyzed (Participants) | 10
Participants | 9

3. Secondary Outcome: Number of Patients With Evidence of Engraftment.
Description: Number of patients who received both cord blood units and achieved sustained donor engraftment
Time Frame: 1 year
Population: 1 patient was not evaluable due to graft failure
Measure: Number; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant Patients
Number analyzed (Participants) | 10
Participants | 2

4. Secondary Outcome: Number of Patients With Acute Graft-versus-host Disease (GVHD)
Description: Number of patients who exhibited grade II-IV acute GVHD at 100 days post umbilical cord blood transplant.
Time Frame: 100 days post transplant
Population: 2 patients were not graded for acute GVHD due to graft failure.
Measure: Number; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant Patients
Number analyzed (Participants) | 8
Participants | 7

5. Secondary Outcome: Number of Patients With Transplant-related Mortality (TRM)
Description: Number of patients who were deceased at days 100 and 180 from any cause other than relapse.
Time Frame: Day 100 and Day 180
Measure: Number; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant Patients
Number analyzed (Participants) | 10
Participants | 5

6. Secondary Outcome: Number of Patients Surviving at Day 100 and 1 Year.
Description: Overall survival of patients-Number of patients who were alive at Day 100 and 1 year post transplant.
Time Frame: Day 100 and 1 year
Measure: Number; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant Patients
Number analyzed (Participants) | 10
Participants | 5

7. Secondary Outcome: Number of Patients With Grade III-IV Acute Graft-versus-host Disease (GVHD)
Description: Number of umbilical cord blood transplant patients developing severe GVHD at 100 days post transplant.
Time Frame: 100 days post transplant
Population: 2 patients were not yet graded for acute gvhd
Measure: Number; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant Patients
Number analyzed (Participants) | 8
Participants | 2

8. Secondary Outcome: Number of Patients With Chronic Graft-versus-host Disease (GVHD).
Description: Number of umbilical cord blood transplant patients with limited and extensive chronic GVHD.
Time Frame: 1 year post transplant
Population: Only 7 patients were at risk for chronic GVHD
Measure: Number; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant Patients
Number analyzed (Participants) | 7
Participants | 2

ADVERSE EVENTS:
Arm/Group | Umbilical Cord Blood Transplant Patients
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umbilical Cord Blood Transplant Patients (N=12)
graft failure (Blood and lymphatic system disorders) | 1 (1)
Acute GVHD Grade 3 (Blood and lymphatic system disorders) | 2 (2)
Death (General disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
This study was terminated early based on interim statistical analysis that indicated time to engraftment will not be improved compared to historical controls. While safe, lack of faster marrow recovery supports early discontinuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No